CLINICAL TRIAL: NCT00236548
Title: An Open-label Evaluation of the Utility of the RISPERDAL CONSTA Treatment Guidebook During Transition of Adult Patients With Schizophrenia or Schizoaffective Disorder to RISPERDAL CONSTA (Risperidone) Treatment Over Three Months in the Community Mental Health Center (CMHC) Setting
Brief Title: Evaluation of the Usefulness to Doctors of the Risperdal Consta Treatment Guidebook Over a Three-month Period During Which Adult Patients With Schizophrenia or Schizoaffective Disorder Are Switching From Daily Doses or Risperidone Tablets to Long-acting Risperidone by Injection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen, LP (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002896
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-03

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Schizophrenia; schizoaffective disorder; patient compliance; long-acting risperidone; intramuscular injection; Treatment Guidebook
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Patient Compliance | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to assess the usefulness of the RisperdalÂ® ConstaÂ® Treatment Guidebook in helping the doctor switch the adult patient from taking risperidone tablets daily by mouth to taking long-acting risperidone by injection. The study will also evaluate the effectiveness and safety of long-acting risperidone and its effect on patient satisfaction.

DETAILED DESCRIPTION:
Many patients who take oral medication to treat schizophrenia or schizoaffective disorder have trouble taking their medication every day. They may not want to take it, or they may just forget. Risperidone injections, given once every 2 weeks, are expected to be just as effective as risperidone tablets taken once a day. The option of getting an injection every 2 weeks rather than taking a tablet every day may help patients keep to their medication administration schedule and could help to reduce the symptoms of their disease. The study will assess the usefulness of the Risperdal® Consta® Treatment Guidebook in a Community Mental Health Center setting, over a period of three months. This Guidebook was designed to help doctors switch adult patients from oral risperidone tablets to long-acting risperidone given once every 2 weeks by injection. During the study, patients will continue to take oral risperidone for 2 weeks following initiation of risperidone injections, which will be given every 2 weeks during a 12-week period. Physical examinations and laboratory tests will be performed to test the safety of the risperidone injections. Both the patient and the doctor will be asked questions about the usefulness of the guidebook and the effectiveness of the injections. The objective of this study is to demonstrate the effectiveness of the Risperdal® Consta™ Treatment Guidebook in switching patients with schizophrenia and schizoaffective disorder from daily oral risperidone to long-acting risperidone injections. In addition, safety evaluations are assessed throughout the study. Risperidone oral tablets, 2 to 6 milligrams per day for the first 2 weeks after initiation of long-acting risperidone injections; long-acting risperidone injections are given in doses of 25, 37.5, or 50 milligrams per 2 milliliter injection once every 2 weeks for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* stable with respect to disease symptoms and other medical conditions
* taking oral risperidone at doses of 2 to 6 milligrams per day for 4 weeks before start of study
* if female, using birth control.

Exclusion Criteria:

* Hospitalized within past 4 weeks to treat exacerbation of symptoms of schizophrenia
* at risk for injury to self or others
* had electroconvulsive therapy within past year
* presence of liver or kidney impairment
* use of oral antipsychotics (other than risperidone) within past 4 weeks, of injected antipsychotics within past 3 months, of clozapine within past 60 days, or of long-acting risperidone in an earlier study
* pregnant or breast-feeding
* not using birth control
* abusing drugs or alcohol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Usefulness of the Risperdal® Consta® Treatment Guidebook; patient and clinician adherence to guidelines

SECONDARY OUTCOMES:
Effectiveness of study drug measured by the Clinical Global Impression scale; safety by assessing treatment-emergent adverse events, vital signs, laboratory tests or electrocardiogram changes; quality of life by the Schizophrenia Quality of Life Scale

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: An open-label evaluation of the RISPERDAL� CONSTA� Treatment Guidebook during transition of adult patients with schizophrenia or schizoaffective disorder to RISPERDAL� CONSTA� over 3 months in the Community Mental Health Center (CMHC) setting — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=499&filename=CR002896_CSR.pdf